CLINICAL TRIAL: NCT03085654
Title: Multiple Dose Effect of Oxytocin on Males With High or Low Trait Anxiety
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UESTC-neuSCAN_10
Record Dates: First submitted 2016-04-15; First posted 2017-03-21 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: multiple doses; oxytocin; trait anxiety

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- High anxiety group (single dose) (Experimental): Oxytocin nasal spray or placebo nasal of one dose in subjects with high trait anxiety.
  Interventions: Drug: Oxytocin nasal spray; Drug: Placebo nasal spray
- High anxiety group (3 doses) (Experimental): Oxytocin nasal spray or placebo nasal spray interleaved during the 5 days( on the 1st,3rd and 5th day),24 IU per day in subjects with high trait anxiety.
  Interventions: Drug: Oxytocin nasal spray; Drug: Placebo nasal spray
- High anxiety group (5 doses) (Experimental): Oxytocin nasal spray or placebo nasal spray for 5 days,24 IU per day in subjects with high trait anxiety.
  Interventions: Drug: Oxytocin nasal spray; Drug: Placebo nasal spray
- Low anxiety group (single dose) (Experimental): Oxytocin nasal spray or placebo nasal spray of one dose in subjects with low trait anxiety.
  Interventions: Drug: Oxytocin nasal spray; Drug: Placebo nasal spray
- Low anxiety group (3 doses) (Experimental): Oxytocin nasal spray or placebo nasal spray interleaved during the 5 days( on the 1st,3rd and 5th day),24 IU per day in subjects with low trait anxiety.
  Interventions: Drug: Oxytocin nasal spray; Drug: Placebo nasal spray
- Low anxiety group (5 doses) (Experimental): Oxytocin nasal spray or placebo nasal spray for 5 days in subjects with low trait anxiety.
  Interventions: Drug: Oxytocin nasal spray; Drug: Placebo nasal spray

INTERVENTIONS:
Drug: Oxytocin nasal spray — Intranasal administration of oxytocin 24 international units per dose.
  Other Names: Oxytocin treatment
Drug: Placebo nasal spray — Intranasal administration of placebo 24 international units per dose.
  Other Names: Placebo control

SUMMARY:
To examine whether multiple doses of oxytocin have different effects on behavior and neural indices in males with high or low trait anxiety.

DETAILED DESCRIPTION:
In the present study, healthy male subjects' trait anxiety levels will be assessed by the sub-trait inventory of the State-Trait Anxiety Inventory (STAI). According to subjects' trait anxiety scores, they will be divided into high or low anxiety experimental groups.

Next, experiments will investigate the acute effect (single dose) and chronic effect (3 doses or 5 doses) of oxytocin on brain functional connectivity during resting-state and brain activation in response to watching emotional stimuli using functional magnetic resonance imaging (fMRI). Also the brain structure data (T1 and diffusion tensor imaging, DTI) of subjects will be collected. After finishing the scanning tasks, subjects will be required to rate the emotional valence, intensity and arousal of the pictures shown in the scanner.

During the course of the study subjects will complete a number of questionnaires: Empathy Quotient (EQ), Cheek and Buss Shyness scale (CBSS),Interpersonal Reactivity Index (IRI),Childhood Trauma Questionnaire (CTQ),Beck depression inventory (BDI), State-Trait Anxiety Inventory (STAI), Autism Spectrum Quotient (ASQ), Liebowitz Social Anxiety Scale (LSAS),Positive and Negative Affect Schedule (PANAS),d2 attention test, and the Visual Analogue Scale for anxiety.

ELIGIBILITY:
Inclusion:

* healthy adult males

Exclusion:

* past or current psychiatric or neurological disorder
* head trauma
* substance abuse
* medication
* fMRI contraindications (e.g. metal implants)

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 147 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Changes between acute and chronic administration of oxytocin on amygdala activity as assessed by fMRI | 5 days
  Changes in neural activity between first dose and repeated dose will be assessed over the time course of 5 days
Changes between acute and chronic administration of oxytocin on amygdala connectivity as assessed by fMRI | 5 days
  Changes in neural connectivity between first dose and repeated dose will be assessed over the time course of 5 days

SECONDARY OUTCOMES:
Interaction of acute and chronic treatment effects with trait anxiety on neural activity | 5 days
  The high and low trait anxiety groups will be compared with respect to differences in the acute effects (single dose, day 1) and changes of effects with chronic treatment over the course of 5 days.
Interaction of acute and chronic treatment effects with trait anxiety on neural connectivity | 5 days
  The high and low trait anxiety groups will be compared with respect to differences in the acute effects (single dose, day 1) and changes of effects with chronic treatment over the course of 5 days.
Effects of oxytocin on arousal ratings of emotional stimuli (acute and changes with chronic treatment) | 5 days
  Subjects will rate arousal of emotional stimuli using Likert Scales
Effects of oxytocin on valence ratings of emotional stimuli (acute and changes with chronic treatment) | 5 days
  Subjects will rate valence of emotional stimuli using Likert Scales
Interaction of treatment effects on valence ratings with trait anxiety (acute and changes with chronic treatment) | 5 days
  The high and low trait anxiety groups will be compared with respect to differences in the acute (single dose, day 1) treatment effects and changes with chronic treatment (5 days)
Interaction of treatment effects on arousal ratings with trait anxiety (acute and changes with chronic treatment) | 5 days
  The high and low trait anxiety groups will be compared with respect to differences in the acute (single dose, day 1) treatment effects and changes with chronic treatment (5 days)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Kendrick, PhD, Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- school of life science and technology, University of Electronic Science and Technology of China, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kou J, Zhang Y, Zhou F, Gao Z, Yao S, Zhao W, Li H, Lei Y, Gao S, Kendrick KM, Becker B. Anxiolytic Effects of Chronic Intranasal Oxytocin on Neural Responses to Threat Are Dose-Frequency Dependent. Psychother Psychosom. 2022;91(4):253-264. doi: 10.1159/000521348. Epub 2022 Jan 27. PMID 35086102